CLINICAL TRIAL: NCT01566864
Title: Multi-Method Health System QI Intervention to Reduce Hypertension Disparities
Brief Title: Multi-Method Health System Quality Improvement Intervention to Reduce Hypertension Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Johns Hopkins Community Physicians (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00037622; 5P50HL105187-02 (NIH)
Record Dates: First submitted 2012-03-22; First posted 2012-03-29 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Hypertension
Keywords: hypertension; disparities; care management; provider education; audit and feedback; Omron; African Americans; organizational change; implementation research
MeSH Terms: conditions — Hypertension | interventions — Ambulatory Care Facilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Behavioral: Improve clinic based measurement of blood pressur (Experimental)
  Interventions: Behavioral: Improve clinic based measurement of blood pressure
- Behavioral: Provider education system to promote patient-cent (Experimental)
  Interventions: Behavioral: Provider education system to promote patient-centered care
- Behavioral: Introduce care management system in clinics (Experimental)
  Interventions: Behavioral: Introduce care management system in clinics

INTERVENTIONS:
Behavioral: Improve clinic based measurement of blood pressure — This intervention seeks to improve BP control and reduce disparities through an organizational change and new skills development. To improve the reliability of BP measurement in clinics, new automated BP machines (Omron HEM-907XL) will be provided for each PCP. Medical assistants will be trained and certified in the proper use of the Omron machine by a master trainer. The will be trained to measure the arm circumference, choose the appropriate cuff and place it properly on the arm. They will be recertified yearly. Once activated, the Omron HEM-907XL will lead measurement for 5 minutes then perform a series of 3 BP measurements spaced by 30 seconds and present the man of these 3 measurements. The mean will be record in the electronic medical records.
  Arms: Behavioral: Improve clinic based measurement of blood pressur
Behavioral: Provider education system to promote patient-centered care — The provider education intervention will address blood pressure control and disparities through audit and feedback. The intervention includes a hypertension dashboard and a linked provider-tailored education intervention. The latter aims to enhance provider communication skills during clinical encounters with hypertension patients, via teaching specific verbal behaviors with practice implications related to elicitation of hypertension treatment and adherence concerns. The dashboard is a web based tool linked to the electronic medical records that imports clinic measurements of BP and offers PCPs a quick assessment of the percentage of those achieving blood pressure control and receiving guideline-concordant care in their panel, clinic, and system overall and by patient race/ethnicity.
  Arms: Behavioral: Provider education system to promote patient-cent
Behavioral: Introduce care management system in clinics — The care management (CM) intervention will address blood pressure management and disparities through patient education, promotion of self-management, and the introduction of an organizational change through the addition of new team members. The CM team will contact patients with a BP of ≥140/≥90 (≥130/≥80 for patients with diabetes mellitus or chronic kidney disease) as identified through the electronic medical records for enrollment in care management services. Patients with a BP in these ranges will be referred to a CM program that emphasizes four key self-management behaviors: diet, physical activity, medication adherence, and self-monitoring. The self-management promotion program will consist of 3 one-on-one sessions either with a Pharm D. or R.D. over the course of 3 months.
  Arms: Behavioral: Introduce care management system in clinics

SUMMARY:
The investigators have designed a three-part quality improvement intervention to 1) improve the clinic-based measurement of blood pressure, 2) introduce a care management system to promote self-management behaviors and rapidly titrate medications by algorithms developed in accord with guidelines and 3) introduce an interactive, needs-based, longitudinal-provider education system that promotes patient-centered care and provides practical examples of patient-provider communication strategies. The intervention will occur at six clinics within the metropolitan area of Baltimore, Maryland. The investigators will also describe clinic and health system characteristics and measure their association with implementation (uptake), success (improvements in blood pressure control and reductions in racial disparities), and sustainability of the three-part intervention over 12 -24 months.

DETAILED DESCRIPTION:
Hypertension is common in the US. From efficacy and observational studies, we know that achieving blood pressure control can reduce morbidity and mortality. However, less than one-third of persons with hypertension achieve control as defined by national guidelines. Furthermore, racial disparities in hypertension have been clearly documented with African American patients being less likely than Caucasians to achieve adequate control. The objective of this study is to study the implementation of a multi-method quality improvement intervention in a pragmatic clinical trial. Six clinic sites within the Johns Hopkins Community Physicians (JHCP) healthcare system have been selected for participation in this study. The sites are located within the metropolitan ara of Baltimore, Maryland, yet differ greatly. We will define the context and local characteristics of each study site and determine which characteristics are associated with blood pressure control and racial disparity at the clinic (micro-system) and health system (macro-system)level. We will deploy a three-part quality improvement intervention to 1) improve the clinic-based measurement of blood pressure, 2) introduce a care management system to promote patients' self-management behaviors and rapidly titrate medications by algorithms developed in accord with guidelines and 3) introduce an interactive, needs-based, longitudinal-provider education system that promotes patient-centered care and provides practical examples of patient-provider communication strategies. Using statistical process control charting, we will determine the stability of blood pressure control in the system prior to intervention and after the introduction of each intervention. We will vary the order of the interventions among the six clinical sites to determine if each intervention is independently effective in each local context and if the effect is repeatable in other contextual situations within the same macro-system. In addition, we will study the organizational characteristics and features of the local context that are associated with implementation, uptake of the interventions and success of each intervention in achieving blood pressure control and reducing racial disparities in blood pressure control at the clinic level .

ELIGIBILITY:
Inclusion Criteria: patients with an ICD9 diagnosis of hypertension or a BP >=120/>=80 who have not been seen in the last 12 months and any patient with their most recent BP >=140/>=90 or >=130/>=80 if they have diabetes mellitus or chronic kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66570 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Percent of clinic patients with controlled blood pressure and the racial disparity in controlled BP at each clinic. | 24 weeks
  The percent of clinic patients each week with SBP < 140 and DBP < 90, or if patient is diabetic or has CKD then SBP <130 and DBP < 80. If no BP measure, patient does not meet JNC-7 guidelines. Note: If multiple BP measures are recorded, the lowest will be used. The racial disparity is defined as the percent difference in blood pressure control between white patients and ethnic minority patients (separated into categories of African-American patients and other race patients). These outcomes will be assessed weekly for 24 weeks prior to and after roll out of each of the interventions.

SECONDARY OUTCOMES:
Terminal digit preference | 24 weeks
  The percent of BP measurements at each clinic that end in zero( or an even number) each week before, during, and after implementation of the BP measurement intervention. The measure will serve as an indicator of the uptake of the OMRON automated BP measurement device. It will be obtained weekly for 24 weeks prior to and after roll out of the BP measurement intervention
Repeat BP measures | 24 weeks
  the percent of patient visits at each clinic each week where a second BP measure was done. This measure will be considered an indicator of the provider's trust of the medical assistant's initial BP recording. The measures will be obtained weekly for 24 weeks prior to and after roll-out of the BP measurement intervention
Patient enrollment in care management | 24 weeks
  The percent of eligible patients who are enrolled in care management with a registered dietitian/pharmacist team. This measurement will be obtained weekly for 24 weeks before and after implementation of the care management intervention.
Completion of care management program | 24 weeks
  Among patients who enroll in care management, the percent of patients who complete 3 intervention contacts with the care management team, The measure will be obtained weekly for 24 weeks before and after implementation of the care management intervention.
Dashboard review/communication skills training completion | 12 months
  The number of dashboard reviews and communication skills training modules completed in each quarter, both divided by the number of providers in each site. This measure will be obtained quarterly for 12 months following the baseline response

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Cooper, MD, MPH, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Community Physicians, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Block L, Flynn SJ, Cooper LA, Lentz C, Hull T, Dietz KB, Boonyasai RT. Promoting sustainability in quality improvement: an evaluation of a web-based continuing education program in blood pressure measurement. BMC Fam Pract. 2018 Jan 10;19(1):13. doi: 10.1186/s12875-017-0682-5. PMID 29320994
- [Derived] Boonyasai RT, Carson KA, Marsteller JA, Dietz KB, Noronha GJ, Hsu YJ, Flynn SJ, Charleston JM, Prokopowicz GP, Miller ER 3rd, Cooper LA. A bundled quality improvement program to standardize clinical blood pressure measurement in primary care. J Clin Hypertens (Greenwich). 2018 Feb;20(2):324-333. doi: 10.1111/jch.13166. Epub 2017 Dec 21. PMID 29267994
- [Derived] Cooper LA, Marsteller JA, Noronha GJ, Flynn SJ, Carson KA, Boonyasai RT, Anderson CA, Aboumatar HJ, Roter DL, Dietz KB, Miller ER 3rd, Prokopowicz GP, Dalcin AT, Charleston JB, Simmons M, Huizinga MM. A multi-level system quality improvement intervention to reduce racial disparities in hypertension care and control: study protocol. Implement Sci. 2013 Jun 4;8:60. doi: 10.1186/1748-5908-8-60. PMID 23734703